CLINICAL TRIAL: NCT01237691
Title: Phase 1 Study of California's HOPE Experiment
Brief Title: An Evaluation of California's Experiment With HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pepperdine University (Other)
Collaborators: University of California, Irvine (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SPPN1110F01
Record Dates: First submitted 2010-11-01; First posted 2010-11-09 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Drugs of Abuse
Keywords: drug use; drug arrests; incarceration
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HOPE supervision (Experimental): Parolee supervised under California's new HOPE parole model.
  Interventions: Behavioral: HOPE supervision
- Parole-as-usual (Active Comparator): Parolees supervised under California parole-as-usual.
  Interventions: Behavioral: Parole-as-usual

INTERVENTIONS:
Behavioral: HOPE supervision — HOPE entails a warning session (Orientation Hearing) where the rules of parole are laid out and parolees are told that any violation of stated parole conditions will be sanctioned with a brief jail term (typically a few days in jail). HOPE includes regular random drug testing.
  Other Names: HOPE; COPE
  Arms: HOPE supervision
Behavioral: Parole-as-usual — Parolees are supervised under standard parole supervision practice in California.
  Other Names: Routine parole
  Arms: Parole-as-usual

SUMMARY:
The phase I evaluation is intended to assess whether or not frequent drug testing and immediate short-term incarceration for drug use and/or other violations and mandated drug treatment for multiple violations, reduces the recurrence of drug use and/or other violation behaviors by California parolees assigned to the study group.

DETAILED DESCRIPTION:
The California HOPE pilot program is being implemented under the authority granted in Penal Code 5058.1. The phase I evaluation is intended to assess whether or not frequent drug testing and immediate short-term incarceration for drug use and/or other violations and mandated drug treatment for multiple violations, reduces the recurrence of drug use and/or other violation behaviors by California parolees assigned to the study group compared with parole-as-usual.

ELIGIBILITY:
Inclusion Criteria:

* Assigned to the Sacramento Metro IV Parole Unit.
* Released from a term of return-to-custody for a violation for, or involving, the use of drugs.
* Have a maximum controlling discharge date at least one year from the date of release from the return-to-custody term.

Exclusion Criteria:

* History of convictions for crimes that require registration under Penal Code Section 290.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2010-11 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Days incarcerated | 24 months
  Total number of days incarcerated in jail or prison

SECONDARY OUTCOMES:
% positive drug tests | 24 months
  Percentage of random and scheduled drug tests that test positive for illicit drugs
%Missed | 24 months
  Percentage of parole appointments that are missed.
Revocation rate | 24 months
  Percentage of parolees that are revoked from probation and returned to prison for either a technical violation or on a new charge.
New arrests | 24 months
  Number of new arrests.
Perceptions of risk of detection | 24 months
  Parolees perceived risk of detection for drug use

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hawken, PhD, Principal Investigator — Pepperdine University
Locations (1):
- Sacramento Metro IV Parole Unit., Sacramento, California, United States